CLINICAL TRIAL: NCT04486716
Title: A Single-arm, Prospective, Multi-center Study to Explore Maintained Efficacy With Ofatumumab Therapy in Patients With Relapsing Multiple Sclerosis Who Discontinue Intravenously Delivered Anti-CD20 Monoclonal Antibody (aCD20 mAb) Therapy (OLIKOS)
Brief Title: A Single Arm Study Evaluating the Efficacy, Safety and Tolerability of Ofatumumab in Patients With Relapsing Multiple Sclerosis
Acronym: OLIKOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GUS07; 111,116 (Other: FDA)
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Ofatumumab; Relapsing multiple sclerosis; MS; RMS; CIS; RRMS; SPM; ocrelizumab; MRI; CD19 B; adult,; OMB157; open-label; rituximab
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Investigational drug will be provided in an autoinjector for subcutaneous administration containing 20 mg ofatumumab (20 mg/0.4 ml) administered at baseline, Day 7, Day 14 and monthly thereafter
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Investigational drug will be provided in an autoinjector for subcutaneous administration containing 20 mg ofatumumab (20 mg/0.4 ml)
  Other Names: OMB157

SUMMARY:
A single arm study evaluating the continued efficacy, safety and tolerability of ofatumumab in patients with relapsing multiple sclerosis who are transitioning from aCD20 mAb therapy

DETAILED DESCRIPTION:
This was a single-arm, multicenter, prospective, study in participants with relapsing multiple sclerosis (MS) who had been previously treated with intravenous (i.v.) anti-CD20 monoclonal antibody (aCD20 mAb) therapy and had received at least 2 consecutive courses of intravenously administered ocrelizumab or rituximab every 6 months, and the last dose was within 4 to 9 months before Baseline/Day 1. In this study, participants could have enrolled only if discontinuing i.v. aCD20 mAb therapy for reasons other than lack of efficacy or due to certain treatment-emergent adverse events (TEAEs). Reasons for switching could have included but were not limited to physician/participant preference, access to commercial drug (e.g. insurance coverage issues), or for other logistical reasons (e.g. geographical relocation, travel, etc.).

Eligible participants received open label ofatumumab 20 mg subcutaneous (s.c.) once monthly for 12 months following initial loading regimen of 20 mg s.c. doses on Days 1, 7, and 14. After the 12-Month Treatment Period there was a Telephone Safety Follow-up call 30 days after last dose of study treatment. The Core phase covered a 28-day Screening Period, 12-Month Treatment Period, and 30-Day Telephone Safety Follow-up.

Upon completing the study, participants could opt to continue ofatumumab therapy through commercial services. Participants who did not continue into the ofatumumab commercial patient services hub within 1 month of the end of study visit or who did not switch to another therapy had to continue into the Post-Treatment Safety Follow-up period, consisting of every 3 month visits including B cell monitoring, until they were able to start on commercial ofatumumab, until they switched to another therapy, or until their B cells were repleted (defined as a B cell concentration greater than the individual participant's baseline value prior to starting the i.v. aCD20 mAb or greater than the lower limit of normal).

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female participants aged 18 to 60 years (inclusive) at screening.
3. Diagnosis of relapsing MS (RMS) according to the 2017 Revised McDonald criteria (Thompson et al. 2018), including CIS, RRMS or SPMS with disease activity as defined by (Lublin et al. 2014).
4. Disability status at Screening with an EDSS score of 0 to 5.5 (inclusive).
5. Received at least 2 courses of intravenous aCD20 mAb (loading doses are considered 1 course):

   • Participants currently treated with ocrelizumab must have received (meet all three criteria below):

1. 2 fully infused initial 300 mg ocrelizumab iv infusions 2. At least 1 fully infused 600 mg ocrelizumab iv infusions 6 months (+/- one month) 3. Last fully infused ocrelizumab dose must have occurred within 4-9 months prior to baseline

•Participants currently treated with rituximab must have received (meet both criteria below):

1. At least 2 fully infused courses of rituximab 500 mg - 1000 mg iv every 6 months (+/- one month).

   1. Initial loading regimens of rituximab i.e. 500 mg - 1000 mg on day 1 and on day 15, are allowed but this is consider a single course and must be followed by additional infusion(s) every 6 months (+/- one month)
2. Last fully infused rituximab dose must have occurred within 4-9 months prior to baseline.

6. Participants discontinuing aCD20 therapy for reasons including, but not limited to: physician/participant preference, access to commercial drug (e.g. insurance coverage issues) or for other logistical reasons (such as geographical relocation, travel, etc.) are eligible for this study. 7. Neurologically stable within 1 month prior to first study drug administration.

8. Must be able to use a smart device or have a caregiver that can assist.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study:

1. Participants that have demonstrated suboptimal response to aCD20 therapy to include:

   a. Signs of MRI activity, defined as ≥ 2 active Gd+ T1 lesions, or any new or newly enlarging T2 lesions, documented within the past 6 months
   * If a prior MRI within the last 6 months is not available, then new or newly enlarging T2 lesions should be considered "not documented" and the patient may continue screening b. Documented relapse while on stable, previous aCD20 treatment.
   * Relapses during the first 3 months of intravenous aCD20 therapy are allowable if the participant is then relapse-free for the 12 months following the relapse while on intravenous aCD20 therapy c. Any signs of clinical worsening as measured by EDSS or any clinical measure documented within the last 6 months
2. Discontinuing aCD20 mAb therapy due to the following treatment- emergent adverse events:

   1. Severe infusion-related reactions (Grade 3 or above)
   2. Recurrent infections defined as ≥ 2 severe infections or ≥ 3 respiratory infections or the need for ≥ 2 courses of antibiotics since starting aCD20 therapy, if the Investigator believes this is related to therapy.
   3. Decreased IgG requiring treatment with Intravenous immunoglobulin
3. Participants with primary progressive MS (Polman et al 2011) or SPMS without disease activity (Lublin et al 2014).
4. Participants meeting criteria for neuromyelitis optica (Wingerchuk et al 2015).
5. Pregnant or nursing (lactating) women
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 6 months after stopping study medication.
7. Participants with active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency).
8. Participants with active systemic bacterial, viral or fungal infections, or known to have acquired immunodeficiency syndrome (AIDS).
9. Participants with neurological symptoms consistent with PML or with confirmed PML.
10. Participants at risk of developing or having reactivation of syphilis or tuberculosis
11. Participants at risk of developing or having reactivation of hepatitis.
12. Have received any live or live-attenuated vaccines (including for varicella-zoster virus or measles) within 4 weeks prior to first study drug administration. a. There is presently no contraindication for the use of an inactivated, viral-vector-or mRNA based Sars-CoV-2 vaccine in patients who are immunocompromised. However, different Sars-CoV-2 vaccines may have various mechanisms of action and different associated potential risks. Please review local prescribing information of any specific Sars-CoV-2 vaccine and comply with local prescribing information requirements for specific contra-indications and special warnings and precautions for use.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - Alabama Neurology Associates PC, Birmingham, Alabama
  - Ctr for Neurology and Spine, Phoenix, Arizona
  - Neuro Center, Pomona, California
  - UC Health Neuroscience Ctr, Aurora, Colorado
  - Infinity Clinical Research LLC, Hollywood, Florida
  - AMO Corporation, Tallahassee, Florida
  - University Of South Florida, Tampa, Florida
  - International Neurorehab Institute, Lutherville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Cente, Boston, Massachusetts
  - Neurology Center of New England PC, Foxborough, Massachusetts
  - Dragonfly Research LLC, Wellesley, Massachusetts
  - Cleveland Clinic Foundation, Las Vegas, Nevada
  - Ms Ctr Of Northeastern Ny, Latham, New York
  - Columbus Neuroscience, Westerville, Ohio
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Parkland Health and Hospital Systems, Dallas, Texas
  - Central TX Neuro Consultants P A, Round Rock, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
- Caribbean Center for Clinical Research, Inc, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Hua LH, Brown B, Camacho E, Chinea AR, Greenberg BM, Henry RG, Houtsma E, Moreo N, Alvarez E. Switch from intravenous anti-CD20 therapy to subcutaneous ofatumumab in patients with relapsing MS: results from the OLIKOS study. J Neurol. 2025 Oct 24;272(11):725. doi: 10.1007/s00415-025-13462-w. PMID 41196386
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is conducted in 20 sites in the United States.
Pre-assignment Details: The study had a Core phase and a Post-Treatment Safety Follow-up (FU). The Core phase covered a 28-day Screening Period, 12-Month Treatment Period, and 30-Day Telephone Safety FU. Upon completing the study, participants could opt to continue ofatumumab therapy through commercial services. Those not continuing with commercial ofatumumab or switching therapies entered the Post-Treatment Safety FU period.
Groups:
- Ofatumumab 20 mg: Subcutaneous injection of ofatumumab 20 mg on Day 1, Day 7, Day 14 and thereafter once monthly starting at Month 1 and up to Month 12.
Period: Core Phase
Arm/Group | Ofatumumab 20 mg
Started (Enrolled participants (completed Screening period)) | 111
Full Analysis Set / Safety Analysis Set (All participants who received at least 1 dose of the study drug) | 102
Completed (Completed study treatment in the Core phase) | 89
Not Completed | 22
Not completed — Subject decision | 6
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Enrolled subjects not treated | 9
Period: Post-Treatment Safety FU
Arm/Group | Ofatumumab 20 mg
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) including all participants who received at least 1 dose of the study drug.
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.51 (8.244)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 78
  Black or African American | 20
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With no Change or a Reduction From Baseline in the Number of Gadolinium Enhancing (GdE) Lesions at Month 12 Using Non-responder Imputation
Description: Magnetic Resonance Imaging (MRI) was used to measure presence of new or reduction in number of gadolinium enhancing T1 lesions. Each MRI scan was previewed by a local neuroradiologist. The quality of each scan performed was assessed by a central MRI reading center and evaluated for quality, completeness and adherence to the protocol.
  A nonresponder imputation (NRI) for missing data approach was applied. NRI assumes that a participant was a treatment failure, i.e. non-responder, if they did not have a valid Month 12 MRI assessment, or if they discontinued the study prematurely and did not have a valid Month 12 MRI assessment.
Time Frame: Baseline (assessed at screening visit), Month 12
Population: Participants in the Full Analysis Set with a value for the outcome measure at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 97
percentage of participants | 86.6 [78.17 to 92.67]

2. Primary Outcome: Percentage of Participants With no Change or a Reduction From Baseline in the Number of Gadolinium Enhancing (GdE) Lesions at Month 12 Based on Observed Data
Description: Magnetic Resonance Imaging (MRI) was used to measure presence of new or reduction in number of gadolinium enhancing T1 lesions. Each MRI scan was previewed by a local neuroradiologist. The quality of each scan performed was assessed by a central MRI reading center and evaluated for quality, completeness and adherence to the protocol.
  A sensitivity analysis of the primary endpoint was performed based on an observed data approach.
Time Frame: Baseline (assessed at screening visit), Month 12
Population: Participants in the Full Analysis Set with a value for the outcome measure at both baseline and Month 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 84
percentage of participants | 100 [95.70 to 100]

3. Secondary Outcome: Number of Participants Who Continued Study Treatment From Baseline to Months 6 and 12
Description: Retention on study treatment from baseline to Month 6 and to Month 12 was based on the number of participants who continued study treatment.
Time Frame: Baseline, Month 6, Month 12
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 102
Participants
  Month 6 | 95
  Month 12 | 89

4. Secondary Outcome: Change From Baseline in CD19+ B Cell Counts Obtained by FACS
Description: Changes from baseline in lymphocytes, including total CD19+ B cell counts and CD20+CD3+ T cell counts, were obtained by fluorescence-activated cell sorting (FACS), which is a specific type of flow cytometry.
Time Frame: Baseline, Month 6, Month 12
Population: Participants in the Safety Analysis Set with an available value for the outcome measure at both baseline and the corresponding time point.
Measure: Mean (Standard Deviation); unit: CD19+ B cells * 10^6/L
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 91
CD19+ B cells * 10^6/L
  Month 6 | -24.45 (58.295)
  Month 12: number analyzed (Participants) | 86
  Month 12 | -17.53 (52.182)

5. Secondary Outcome: Change From Baseline in CD20+ CD3+ T Cell Counts Obtained by FACS
Description: as for outcome 4
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: CD20+ CD3+ T cells * 10^6/L
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 88
CD20+ CD3+ T cells * 10^6/L
  Month 6 | -11.144 (39.1520)
  Month 12: number analyzed (Participants) | 77
  Month 12 | -2.590 (32.1112)

6. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire that assesses suicidal ideation and suicidal behavior. The suicidal ideation section includes 5 items (Categories 1 to 5), and the suicidal behavior section includes 5 items (Categories 6 to 10). Additionally, there is one item about Self-injurious behavior, without suicidal intent.
  The C-SSRS was given multiple times throughout the study from baseline up to Month 12. The number of participants who answered 'Yes' to any of the items in C-SSRS at baseline and at any timepoint post-baseline is summarized in this record.
  Baseline refers to all prior history.
Time Frame: Baseline (all prior history), Post-baseline (up to Month 12)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 102
Participants
  Baseline: Any suicidal ideation (Categories 1 to 5) | 18
  Baseline: Any suicidal behavior (Categories 6 to 10) | 6
  Baseline: Any suicidal ideation or behavior (Categories 1 to 10) | 19
  Baseline: Self-injurious behavior, without suicidal intent | 4
  Post-baseline: Any suicidal ideation (Categories 1 to 5) | 4
  Post-baseline: Any suicidal behavior (Categories 6 to 10) | 0
  Post-baseline: Any suicidal ideation or behavior (Categories 1 to 10) | 4
  Post-baseline: Self-injurious behavior, without suicidal intent | 0

7. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) Scores at Baseline, Month 6 and Month 12
Description: The Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) is a 9-item general instrument that measures the major dimensions of satisfaction with a medication. The questionnaire consists of 3 domains: effectiveness (items 1 to 3), convenience (items 4 to 6) and global satisfaction (items 7 to 9). The scores of each domain range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Time Frame: Baseline, Month 6, Month 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at each time point.
Measure: Median (Full Range); unit: Score on scale
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 51
Score on scale
  TSQM-9 Effectiveness Score - Baseline | 61.11 [0.0 to 100.0]
  TSQM-9 Effectiveness Score - Month 6: number analyzed (Participants) | 41
  TSQM-9 Effectiveness Score - Month 6 | 66.67 [5.6 to 100.0]
  TSQM-9 Effectiveness Score - Month 12: number analyzed (Participants) | 42
  TSQM-9 Effectiveness Score - Month 12 | 66.67 [11.1 to 100.0]
  TSQM-9 Convenience Score - Baseline | 61.11 [22.2 to 100.0]
  TSQM-9 Convenience Score - Month 6: number analyzed (Participants) | 41
  TSQM-9 Convenience Score - Month 6 | 88.89 [50.0 to 100.0]
  TSQM-9 Convenience Score - Month 12: number analyzed (Participants) | 42
  TSQM-9 Convenience Score - Month 12 | 86.11 [50.0 to 100.0]
  TSQM-9 Global Satisfaction Score - Baseline | 63.89 [5.6 to 100.0]
  TSQM-9 Global Satisfaction Score - Month 6: number analyzed (Participants) | 41
  TSQM-9 Global Satisfaction Score - Month 6 | 77.78 [33.3 to 100.0]
  TSQM-9 Global Satisfaction Score - Month 12: number analyzed (Participants) | 42
  TSQM-9 Global Satisfaction Score - Month 12 | 42.22 [33.3 to 100.0]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any adverse events (AEs) that started on or after the day of first dose of study drug, or before 30 days after the treatment end date, if severity at baseline was missing or if postbaseline severity was greater than baseline severity.
Time Frame: From first dose of study drug (Day 1) up to 30 days after last dose (Month 13)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab 20 mg
Number analyzed (Participants) | 102
Participants
  Participants with AEs (any AE, regardless of seriousness) | 86
  Participants with serious adverse events (SAEs) | 6

ADVERSE EVENTS:
Time Frame: From first dose (Day 1) through the safety follow-up period, with an average duration of 30 days after last dose (approximately 13 months total) and a maximum follow-up of up to 18 months post-dose (approximately 30 months total).
Arm/Group | Ofatumumab 20 mg
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 6/102
Other Adverse Events (participants affected / at risk) | 53/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 20 mg (N=102)
COVID-19 (Infections and infestations) | 1
Infective myositis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Sciatic nerve injury (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 20 mg (N=102)
Fatigue (General disorders and administration site conditions) | 12
Pyrexia (General disorders and administration site conditions) | 6
COVID-19 (Infections and infestations) | 31
Urinary tract infection (Infections and infestations) | 11
Headache (Nervous system disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT04486716/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04486716/SAP_001.pdf